CLINICAL TRIAL: NCT03517475
Title: Prevention of Injuries Among Young Children: Tailoring a Home Supervision Intervention for Low-Income Caregivers
Brief Title: Tailoring a Home Supervision Intervention for Low-Income Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Collaborators: University of Guelph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AD3874920
Record Dates: First submitted 2018-02-26; First posted 2018-05-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervising for Home Safety modified (Experimental): We will train caregivers to provide adequate levels of supervision to the 3-4 year-old children.
  Interventions: Behavioral: SHS Low-Income
- Services as Usual (Placebo Comparator): Clients will receive home visiting services from Head Start
  Interventions: Behavioral: SHS Low-Income

INTERVENTIONS:
Behavioral: SHS Low-Income — An intervention to train caregivers to supervise their children appropriately.

SUMMARY:
The investigators will pilot test (N=100 caregivers of children ages 3-4 years) the effects of a caregiver supervision intervention on caregivers' supervision and children's injury frequency using a Randomized Controlled Trial (RCT) design. The control group will receive Services as Usual (SAU), and the treatment group will receive SAU+ SHS. The results will be used to support an R01 application to conduct a larger-scale RCT test of the program.

DETAILED DESCRIPTION:
For the RCT, the investigators will recruit Head Start participants with help from the home visitors (using procedures that are similar to phase 1 recruitment procedures). The home visitors will read a short script about the study to eligible clients; it will be emphasized that the Head Start services they receive will not be impacted by their decision about whether or not to participate. Interested caregivers will sign a release form for the home visitors to provide the caregiver's contact information to study personnel. A Graduate Research Assistant (GRA) will then call the caregivers and will read a recruitment script. If the caregiver is interested in participating, the GRA will set up a meeting in the caregiver's home to complete consent and baseline measures. Caregivers will be eligible to participate if they are the primary caregiver (male or female) for at least one child in the target age range (3-4 years-of-age), the caregiver can speak and read English, and the caregiver did not participate in the focus group study. The investigators will exclude families in which the target child has been diagnosed with a pervasive developmental disorder or is blind or deaf because such conditions often result in specialized supervision requirements, and the investigators have not tailored the intervention to be appropriate for such families. Later research may examine whether the intervention or a modified version of it, is appropriate for such families. If there is more than one child in the home who is attending Head Start and is between the ages of 3-4 years, the investigators will use a random procedure to choose the target child. Participants who consent will be randomly assigned to either the treatment or control condition by the primary investigator after the consent appointment. A blinded design will be used so the GRA who will collect data will not know who is in the treatment group.

A GRA and URA will administer baseline, post-test, and follow-up assessments at participants' homes. Baseline assessments will include three self-report measures of caregiver supervision beliefs and practices, a measure of caregivers' injury beliefs, and a measure of children's injury history. The investigators will also conduct an observation of in-home supervision and collect data on current injuries. The baseline, post, and follow-up sessions will take approximately one hour. If needed, the GRA will assist caregivers with low literacy to complete the measures by reading the measures aloud or by answering questions about the measures. The investigators have used this approach successfully in previous studies (Damashek & Corlis, 2017; Damashek, Hughes, Chahin, & Corlis, 2017). After the baseline session, primary caregivers randomized to the treatment condition will participate in one-hour intervention sessions in their home for 5 weeks. Those randomized to the treatment group will receive the tailored SHS intervention in addition to their Head Start home visiting services (SHS+SAU); those randomized to the control group will only receive the Head Start home visiting services (SAU). A GRA will deliver the intervention to the treatment group and will be assisted by an Undergraduate Research Assistant (URA). The GRA will be trained by the co-investigator to deliver SHS and will use a manual to guide delivery (based on previous work, Morrongiello et al., 2017).

A week after the last intervention session (or an equivalent time period for the control group), the GRA and URA will return to the participant's home and will re-administer the same measures taken at baseline, in addition to questionnaires assessing their satisfaction with the intervention and perception of the intervention's cultural acceptability. The investigators will conduct a 1-month follow-up to assess for sustainability of effects during which the investigators will administer the same supervision and injury measures as at baseline.

In addition to self-report measures, the investigators will conduct pre-, post-, and follow-up observational assessments of maternal supervision, based on an innovative testing protocol developed by Morrongiello and her colleagues (Morrongiello, McArthur, Goodman, & Bell, 2015). During the data collection appointments, the investigators will set up a situation in which the investigators will observe caregivers' supervision of their child while they are distracted and while their child is exposed to an interesting and potentially hazardous object (a "gadget", see Measures).

The investigators will also collect data on children's minor everyday injury frequencies using a structured injury interview that will be administered weekly via telephone; this measure has been used in previous research by the PI (Damashek & Corlis, 2017). The first interview will be administered in person during the baseline data collection session. A second baseline injury interview will occur 1 week before caregivers participate in their first intervention session. Additional administrations will occur weekly via telephone through the follow-up data collection appointment.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers will be eligible to participate if they are the primary caregiver (male or female) for at least one child in the target age range (3-4 years-of-age), the caregiver can speak and read English, and the caregiver did not participate in the focus group study.

Exclusion Criteria:

* We will exclude families in which the target child has been diagnosed with a pervasive developmental disorder or is blind or deaf.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Supervision levels | 11 weeks

SECONDARY OUTCOMES:
Injury Frequency | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy Damashek, Principal Investigator — Western Michigan University
Locations (1):
- Western Michigan University, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided